CLINICAL TRIAL: NCT00702364
Title: Strattera(Atomoxetine) for the Treatment of Attention Disorders in Individuals With Traumatic Brain Injury
Brief Title: Efficacy Study of Strattera for Treating Attention Disorders in Traumatic Brain Injury (TBI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Craig Hospital (Other)
Responsible Party: Principal Investigator, Cynthia Harrison-Felix, PhD, Assistant Director of Research, Craig Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H133A07022R01
Record Dates: First submitted 2008-06-18; First posted 2008-06-20 (Estimated); Results first posted 2014-09-15 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-08

CONDITIONS: Traumatic Brain INjury
Keywords: Attention; Traumatic Brain INjury; Atomoxetine; Strattera
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atomoxetine (Experimental): 40mg atomoxetine twice a day for 2 weeks
  Interventions: Drug: atomoxetine
- placebo (Placebo Comparator): Placebo twice a day for two weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: atomoxetine
  Other Names: strattera
  Arms: Atomoxetine
Drug: placebo
  Arms: placebo

SUMMARY:
Atomoxetine is the only medication that is currently approved by the FDA for the treatment of attention deficit hyperactivity disorder in adults. It has gained recent interest as an alternative medication for treating attentional problems related to traumatic brain injury (TBI), but it's effectiveness in this population has not been studied. There are a number of advantages of Atomoxetine over traditional neuro-stimulant medications currently used for attentional disorders after traumatic brain injury. This study will use a randomized double-blind placebo-controlled crossover design to investigate the efficacy of atomoxetine to improve attention, behavioral function, and depression in adults with TBI

ELIGIBILITY:
Inclusion Criteria:

* History of TBI
* Moderate to severe TBI as indicated by Glasgow Coma Score (GCS) score of 12 or less; or Post Traumatic Amnesia (PTA) of seven days or more
* at least one year post injury
* between the ages of 18-65 (inclusive)
* symptoms consistent with attentional dysfunction
* consent to participate in study

Exclusion Criteria:

* history of any conditions that would prohibit standard neuropsychological testing
* non-English speaking (to the extent that would limit ability to complete study measures)
* prior history of significant psychiatric illness requiring hospitalization
* epilepsy
* cardiovascular disease or risks including: dysrhythmias, angina, myocardial infarction, uncontrolled hypertension, valvular heart disease including mitral valve prolapse
* use of any monoamine oxidase inhibitor or any other drug affecting brain monoamine concentrations
* severe renal or hepatic impairment
* pregnant or lactating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David L Ripley, MD, Principal Investigator — Craig Hospital; Cindy Harrison-Felix, PhD, Principal Investigator — Craig Hospital
Locations (1):
- Craig Hospital, Englewood, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 175 people responded to recruitment flier in the Denver area and were screened for eligibility from April 2008 through December 2011. 60 of these enrolled in the study.
Pre-assignment Details: 60 enrolled participants completed study training; 2 of these withdrew prior to Baseline Assessment. 58 completed baseline assessment and began Placebo Run-in; 3 withdrew prior to randomization. 55 total were randomized.
Groups:
- Atomoxetine: 40mg atomoxetine twice a day for 2 weeks
  atomoxetine :
- Placebo: Placebo twice a day for two weeks
  placebo :
Period: Overall Study
Arm/Group | Atomoxetine | Placebo
Started | 26 | 29
Completed | 24 | 25
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Population: Baseline analysis was completed on the 55 randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Atomoxetine | Placebo | Total
Number analyzed (Participants) | 26 | 29 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 29 | 55
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 18 | 23 | 41

OUTCOME MEASURES:

1. Primary Outcome: CDR Power of Attention
Description: Cognitive Drug Research (CDR) Computerized Cognitive Assessment System [19] is comprised of a battery of computer-controlled tasks administered on a laptop computer with parallel forms of the tests being presented on each testing session. The Power of Attention factor of the CDR was selected as the primary outcome measure because of its strong psychometric properties in other drug studies with cognitively compromised populations.
  Instead of utilizing a t-test to compare treatment and control groups, treatment and control groups for both primary and secondary outcomes were compared utilizing an analysis of covariance (ANCOVA) model in which repeat baseline measures taken on each respective outcome served as a covariate. This method controls for any differences that may exist between the groups at baseline. Model assumptions for conducting an ANCOVA were investigated for all primary and secondary analyses, where no violations of model assumptions were detected. Additionally,
Time Frame: Post treatment
Measure: Mean (95% Confidence Interval); unit: msec
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 25 | 28
msec | 1262.1744 [1209.8949 to 1314.4539] | 1252.9510 [1203.6002 to 1302.3019]

2. Primary Outcome: Stroop Test Interference T-score
Description: The Stroop Color and Word Test is frequently used to study deficits of attention and executive function in individuals with TBI, and has adequate test-retest reliability. At each administration, the following scores were obtained, Word Reading, Colour Naming and Interference. Raw scores were converted to demographically-adjusted T-scores using Golden and Freshwater norm.
Time Frame: Post treatment
Measure: Mean (95% Confidence Interval); unit: T-score
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 25 | 28
T-score | 56.50 [54.70 to 58.30] | 55.44 [53.74 to 57.14]

3. Primary Outcome: Adult Attention Deficit Hyperactivity Disorder (ADHD) Self-Report Scale Summary Score
Description: The Adult ADHD Self-Report Scale (ASRS-v1.1) is a self-report questionnaire that consists of questions involving the 18-items of the The Diagnostic and Statistical Manual of Mental Disorders (DSM)-IV- Text Revision (TR) criteria for ADHD that rate symptoms on a Likert scale ranging from 0-4 based on the frequency of symptoms ("never", "rarely", "sometimes", "often", and "very often"). A previous study of the ASRS found the self-report to be both valid (Cronbach's alpha =.88) and reliable (ICC=.84). Scores on the 18 items were summed for a total ASRS score.
Time Frame: Post treatment
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 25 | 28
units on a scale | 28.883 [25.746 to 32.021] | 30.997 [28.033 to 33.959]

4. Secondary Outcome: Neurobehavioral Functioning Inventory Depression Subscale
Description: Neurobehavioral Functioning Inventory (NFI) was developed as a clinical and research tool to quantify a variety of post-injury behaviours and symptoms characteristic of neurologic disability and encountered in daily life. The inventory is comprised of 76 items organized into six analytically derived factor scales: Depression, Somatic, Memory/Attention, Communication, Aggression, and Motor. Respondents are asked to rate items as occurring "never", "rarely", "sometimes", "often", or "always". Using the standardized scoring procedures outlined in the NFI Manual, T-scores were calculated for the Depression sub-scale. Lower T-score indicates less depressive symptomotology.
Time Frame: Post treatment
Measure: Mean (95% Confidence Interval); unit: T-score
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 25 | 28
T-score | 27.53 [24.87 to 30.18] | 29.47 [26.92 to 32.02]

ADVERSE EVENTS:
Arm/Group | Atomoxetine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/29
Other Adverse Events (participants affected / at risk) | 0/26 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes